CLINICAL TRIAL: NCT00510172
Title: Migraine Inducing Effects and Changes in Brain Haemodynamics of PGI2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: KA-20060086
Record Dates: First submitted 2007-07-30; First posted 2007-08-01 (Estimated); Last update posted 2007-08-01 (Estimated); Status verified 2007-07

CONDITIONS: Headache; Migraine; Vasodilatation
Keywords: Headache; Migraine; Vasodilatation
MeSH Terms: conditions — Headache; Migraine Disorders; Aneurysm | interventions — Epoprostenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Active treatment
  Interventions: Drug: Prostacyclin, PGI2
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prostacyclin, PGI2 — 10 ng/kg/min of epoprostenol (stable PGI2)
  Arms: 1
Drug: Placebo — NaCL 0,9%
  Arms: 2

SUMMARY:
We hypothesised that intravenous infusion of PGI2 induced headache or migraine and cranial vasodilatation in migraineurs.

ELIGIBILITY:
Inclusion Criteria:

* migraine without aura and healthy apart from that
* age 18-55 years
* 50-100 kg
* Secure contraceptives

Exclusion Criteria:

* Tension Type Headache more than 3 time a month
* Other primary headaches
* Medication prior to the study (closer than 4 times plasma halflife)
* Migraine or headache 5 days prior to study.
* Hypertension (systolic BP >150 mmHg and/or diastolic BP >100 mmHg).
* Hypotension (systolic BP <90 mmHg and/or diastolic BP <50 mmHg).
* Heart-vessel disease of any kind incl cerebrovascular disease.
* Anamnestic or clinical signs of psychiatric disease or abuse.
* Anamnestic or clinical signs of disease of any kind relevant for participation in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2006-12; Study Completion 2007-09 (Estimated)

PRIMARY OUTCOMES:
Headache and accompanying symptoms. Blood flow velocity in the middle cerebral artery, diameter changes in superficial temporal artery and radial artery. | 14 hours

SECONDARY OUTCOMES:
Blood pressure, pulse | 100 min

CONTACTS AND LOCATIONS:
Overall Officials: Troels Wienecke, MD, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Copenhagen, Glostrup, Denmark